CLINICAL TRIAL: NCT01782716
Title: Effect of Different Scoring Systems on Mortality Rates and Length of Hospitalization in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Cumhuriyet University Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Cemil Isbir, M.D, Cumhuriyet University
Other Study IDs: Other Identifier-2011/037
Record Dates: First submitted 2013-01-30; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2011-12

CONDITIONS: Heart Diseases
Keywords: Mortality; Length; hospitalization; cardiac surgery; patients
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ASA
- ASA+Euroscore

SUMMARY:
Precise risk estimation of mortality in cardiac surgery patients is often difficult. Main objectives of this study is to calculate mortality probability by two different risk score system and to inquire effects of informing anesthesiologist and surgical team; of score of the patient; on length of hospitalization and intensive care and also on actualized mortality.

ELIGIBILITY:
Inclusion Criteria:

* ASA anesthesia risk group 2-5 patients between 18-70 years of age and with planned cardiac surgery

Exclusion Criteria:

* Terminal malignant diagnosis, multiple organ failure, confirmed brain dead, mechanical ventilation dependent or planned transplantation patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery patients
Sampling Method: Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The number of days the patients treated | 30 days
mortality | With in the 30 days after surgery